CLINICAL TRIAL: NCT04126694
Title: Using Continuous Glucose Monitoring to Detect and Intervene on Maintenance Factors for Trans-diagnostic Binge Eating Pathology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1907007293
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Bulimia Nervosa; Binge Eating
MeSH Terms: conditions — Bulimia Nervosa; Bulimia

STUDY DESIGN:
Intervention Model Description: Participants will receive 12 sessions of in-person CBT delivered over 12 weeks. In weeks 1-2, participants will wear the CGM devices, but will not receive JITAIs and therapists will not have access to the clinician portal. During weeks 3-4, JITAIs will be "turned on" such that patients begin to receive push notifications based on CGM data and therapists will have access to the clinician portal. The A/B periods will be repeated (weeks 5-6 and 9-10, SenseSupport Off; weeks 7-8 and 11-12 SenseSupport On) to ensure that improvements in dietary restriction are due to SenseSupport and not simply to the effect of time in treatment. Similar to the approach used in prior studies, participants will be ran in small waves (n= 3-5 per wave). During each wave, feasibility, acceptability, and target engagement will be assessed, and if acceptable milestones have not been achieved, SenseSupport will be modified before beginning the next wave.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBT with smartphone application (Experimental): 12 weeks of CBT with SenseSupport smartphone application
  Interventions: Behavioral: CBT with smartphone application SenseSupport

INTERVENTIONS:
Behavioral: CBT with smartphone application SenseSupport — SenseSupport intervention system used as an augment to a 12 week in-person CBT treatment for transdiagnostic binge eating pathology

SUMMARY:
The current study will be one of the first to develop and test a passive data collection technique to detect both meal consumption and disordered eating symptoms in patients with clinically significant binge eating and the first just-in-time adaptive interventions (JITAIs) systems using passive sensing technology for eating pathology to be empirically evaluated. A small iterative open clinical trial using an ABAB design (A= SenseSupport Off, B=SenseSupport On) will be conducted to test the feasibility, acceptability, and target engagement of SenseSupport when paired with a 12 week in-person CBT treatment program. The hypothesis that larger decreases in dietary restriction will be observed during SenseSupport On phases compared to SenseSupport Off phases will be tested in this clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 to 65 years old
* Experience clinically significant binge eating (defined as 12 or more objectively large binge eating episodes in the past 3 months)
* Engage in clinically significant dietary restriction (define as >1 standard deviation above community norms on the Eating Disorder Examination Dietary Restraint Subscale)
* Have a BMI above 18.5
* Are able to give consent

Exclusion Criteria:

* Are unable to fluently speak, write and read English
* Are receiving treatment for an eating disorder
* Require immediate treatment for medical complications as a result of eating disorder symptoms
* Have a mental handicap, or are experiencing other severe psychopathology that would limit the participants' ability to comply with the demands of the current study (e.g. severe depression with suicidal intent, active psychotic disorder)
* Have diabetes
* Are pregnant or planning to become pregnant within the next year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Number of weekly episodes of going ≥ 4 waking hours without eating | 12 weeks
  The number of weekly episodes of going ≥ 4 waking hours without eating captured through CGM and EMA data as well as an EDE-Q assessment before each weekly therapy session. Higher numbers indicate more weekly episodes of dietary restriction. There are no subscale scores or a total score. The number of weekly episodes of going ≥ 4 waking hours without eating will be used to assess the amount of dietary restriction occurring throughout the course of treatment as compared to baseline dietary restriction for the participant.

SECONDARY OUTCOMES:
Eating Disorder Examination Questionnaire (EDE-Q) | Assessed before each weekly treatment session throughout treatment duration (12 weeks)
  The Eating Disorder Examination Questionnaire measures eating pathology. The EDE-Q yields four subscale scores: Restraint, Eating Concern, Shape Concern, and Weight Concern. The possible score range for each subscale is 0 to 6. The total score may also be reported (determined by averaging the subscale scores); the score range for the total score is also 0 to 6. For subscale scores and total score, higher scores indicate more severe pathology. The restraint sub-scale of the EDE-Q will be used to assess utilization of skills related to reducing dietary restraint.
Feedback Questionnaire (FQ) | Assessed at weekly treatment sessions throughout treatment duration (12 weeks)
  The feedback questionnaire asks qualitative questions about the application. The feedback questionnaire does not report either subscale scores or a total score. The FQ will be used to obtain qualitative acceptability ratings.
Technology Acceptance Model Scale (TAMS) | Assessed at weekly treatment sessions throughout treatment duration (12 weeks)
  The Technology Acceptance Model Scale measures usefulness and ease of use of a technological product. The TAMS yields two subscale scores (usefulness and ease of use). The possible score range for each subscale is 6 to 49. Higher scores indicate greater usefulness and ease of use. The TAMS will be used to assess the perceived usefulness and perceived ease-of-use of the smartphone application to evaluate acceptability.

CONTACTS AND LOCATIONS:
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Juarascio AS, Srivastava P, Presseller EK, Lin M, Patarinski AGG, Manasse SM, Forman EM. Using Continuous Glucose Monitoring to Detect and Intervene on Dietary Restriction in Individuals With Binge Eating: The SenseSupport Withdrawal Design Study. JMIR Form Res. 2022 Dec 14;6(12):e38479. doi: 10.2196/38479. PMID 36515992